CLINICAL TRIAL: NCT07184190
Title: Effects of Trancutaneous Auriculotemporal Nerve Stimulation on Nociceptive Processing. A Randomized, Double-blind, Crossover Pilot Clinical Trial.
Brief Title: Effects of Trancutaneous Auriculotemporal Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Mauro Barone, Principal Investigator, University of Gran Rosario
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25/20
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Neuromodulation; Transcutaneous nerve stimulation; Pressure Pain Threshold; Temporal Summation of Pain; Conditioned Pain Modulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Auriculotemporal Nerve Stimulation (TENS) (Experimental): The tANS (TENS) will be administered using clip electrodes placed on the auricular helix for 30 minutes per session. Stimulation parameters will be: alternating frequency to avoid tolerance; low frequency (2-10 Hz); and high frequency (50-100 Hz). The pulse width will be 125-200 μs, and the current intensity will be individually adjusted to produce a strong but non-painful sensory response.
  Interventions: Other: Trancutaneous Auriculotemporal Nerve Stimulation
- Transcutaneous Auriculotemporal Nerve Stimulation (EE) (Active Comparator): The tANS (EE) will be administered using clip electrodes placed on the auricular helix for 30 minutes per session. Stimulation parameters will be: biphasic rectangular pulses, with a frequency between 30 and 60 Hz, a pulse width of 200 to 300 μs, a 20-second on / 20-second off duty cycle, and a 2-second ramp-up and ramp-down phase. The current intensity will be individually adjusted to produce a strong but non-painful sensory response.
  Interventions: Other: Trancutaneous Auriculotemporal Nerve Stimulation

INTERVENTIONS:
Other: Trancutaneous Auriculotemporal Nerve Stimulation — Trancutaneous Auriculotemporal Nerve Stimulation

SUMMARY:
Neuromodulation works by either actively stimulating nerves, causing the alteration or modulation of nerve activity by delivering electrical agents directly to a target area.

Transcutaneous auricular vagus nerve stimulation is a noninvasive therapy that has demonstrated positive effects in a wide range of conditions. The auricular branch of the vagus nerve is stimulated by electrical pulses in the skin of the ear (cymba conchae). Knowledge about the effects of trigeminal nerve stimulation has increased considerably in recent decades, demonstrating great potential as a therapeutic tool. However, to date, no studies have evaluated the effects of transcutaneous auriculotemporal nerve stimulation (tANS).

Therefore, the aim of this study will be to compare the effects of two types of tANS on nociceptive processing in asymptomatic volunteers.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, crossover pilot clinical trial. Its objective is to compare the immediate effects of two types of transcutaneous auriculotemporal nerve stimulation (tANS) applied to the auricular helix on nociceptive processing in asymptomatic volunteers.

Outcome measures will include pressure pain threshold, temporal summation of pain, and conditioned pain modulation. Adverse effects and treatment tolerance will also be recorded.

Eligible participants will be randomly assigned to one of two groups:

Group 1: tANS using transcutaneous electrical nerve stimulation (TENS)

Group 2: tANS using electrical stimulation (ES)

Each intervention will be administered 72 hours apart at the University of Greater Rosario (Rosario, Argentina).

Outcomes will be assessed both before and after each treatment. All assessments will be conducted by a physical therapist blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes, aged 18 to 35 years;
* No symptoms or history of disease in the craniofacial region;
* No symptoms of chronic pain in any body region.

Exclusion Criteria:

* History of surgery, trauma to the craniofacial region or cancer;
* Systemic disease (e.g., rheumatic disease);
* Neurological and/or psychiatric disorders;
* Altered sensation (e.g., hipo or hypersensitivity);
* Current pregnancy or menstrual cycle
* Intake medication (e.g., centrally acting);
* Prior experience with electrical stimulation treatment;
* Intense physical activity, use of stimulants and/or analgesics in the previous 24 hours;
* Acute sleep disruptions (e.g., recent sleep deprivation);
* Inability to understand the informed consent document.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
1. Change in Pressure Pain Threshold | Pre-intervention and post-intervention with a 72 hours washout period, between groups
  The Pressure Pain Threshold (PPT) will be measured through a pressure algometer in 2 different sites bilaterally; 1) temporomandibular joint and 2) thenar eminence. At each site, 3 measurements will be made with an interval of 30 seconds, and the mean will be registered. To determine the PPT, the pressure will be increased at a rate of approximately 1 kg/second and patients will be asked to raise their arm the moment the pressure begins to change to a sensation of pain, at which point, the evaluator will stop pressing. PPT values will be expressed in kg/cm2. The PPT will be determined as the arithmetic mean of the three measurements. A higher score means a better result.
Change in Temporal Summation of Pain | Pre-intervention and post-intervention with a 72 hours washout period, between groups
  Temporal Summation of Pain (TSP) will be induced using a pressure algometer. For TSP, 10 consecutive pressure pulses will be elicited using the PPT (obtained before). For each pulse of the TSP procedure, the pressure will increase at a rate of 1 kg/second until the PPT is reached, where it will remain for one second before being released. The pressure pulses will be repeatedly performed with an interval between stimuli of one second. Participants will be instructed to assess the pain intensity of the first and tenth pressure pulses according to the numeric pain rating scale (NPRS). The TSP score will be obtained by subtracting the first NPRS score from the last score. The higher the TSP score, the more efficient the nociceptive signaling for the brain.
Change in Conditioned Pain Modulation | Pre-intervention and post-intervention with a 72 hours washout period, between groups
  For Conditioned Pain Modulation (CPM), cold water immersion will be used as the conditioning stimulus (CS) and the PPT as the test stimulus (TS). The participant will immerse their non-dominant hand in a cold water bath at approximately 4°C (±0.5°C) until they reach their maximum pain tolerance or 2 minutes after the start of the immersion, at which point they will remove their hand. The TS will be taken before and immediately after the CS (three PPT measurements). Differences between the PPT values before and after the CS will be considered as CPM values. A greater difference in score indicates more efficient descending inhibition.

SECONDARY OUTCOMES:
Adverse Effects And Tolerance | Time Frame: Immediately and 72 hours after the interventions.
  Participants will be asked about the presence of adverse effects immediately and 72 hours after the stimulations (e.g., itching or skin irritability at the electrode placement site) and their assessment of which stimulation was best tolerated (using the numerical pain rating scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad del Gran Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
The information shared, if required, will be the Statistical Analysis Plan and Informed Consent Form.
Supporting Information: SAP, ICF